CLINICAL TRIAL: NCT07169708
Title: A Retrospective Observational Study of Nivolumab in Combination With Chemotherapy as Neoadjuvant Therapy for Resectable NSCLC Patients: Real-World Experience in Taiwan
Brief Title: A Retrospective Observational Study of Nivolumab in Combination With Chemotherapy as Neoadjuvant Therapy for Resectable NSCLC Patients: Real-World Experience in Taiwan (NEOREAL)
Status: Not yet recruiting | Type: Observational
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: R1132-NIV-24
Record Dates: First submitted 2025-08-28; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-07

CONDITIONS: Non Small Cell Lung Cancer NSCLC
Keywords: NeoReal; NSCLC; Nivolumab; Opdivo; Neoadjuvant therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Resectable NSCLC Patients: Receive Nivolumab in Combination with Chemotherapy

SUMMARY:
The goal of this observational study is to learn about the effectiveness of Nivolumab in combination with chemotherapy as Neoadjuvant therapy for patients with non-small cell lung cancer (NSCLC). The main question it aims to answer is:

Does patient with NSCLC in treatment of Nivolumab combined with chemotherapy demonstrate better pCR and PFS ? Is it safe for patient with NSCLC in treatment of Nivolumab combined with chemotherapy ?

The data for those participants already receiving nivolumab in combination with chemotherapy as part of their regular medical care for NSCLC will be collected within the designated collection period.

DETAILED DESCRIPTION:
Rationale :

In Taiwan, lung cancer is the most common cancer and has the highest mortality rate among the top 10 cancers, accounting for 19.4% of all cancer-related deaths in 2022. Additionally, 94.3% of lung cancer cases were diagnosed as NSCLC (n = 16,420). Based on clinical staging (per AJCC 8th edition), 2.26% of NSCLC cases were classified as stage 0, 35.75% as stage I, 3.79% as stage II, 8.80% as stage III, 41.01% as stage IV, and 8.39% had an unknown stage.25 The US Food and Drug Administration (FDA) approved nivolumab in combination with platinum-doublet chemotherapy for the neoadjuvant treatment of patients with resectable NSCLC in March 2022 and Taiwan subsequently approved this indication in February 2023. However, the real-world effectiveness of this treatment and the NSCLC patient profile, particularly in the Taiwanese population, remains unclear, as does the patient profile for adjuvant therapy following neoadjuvant chemo-immunotherapy (chemo-IO). Therefore, this study aims to address these gaps and consolidate nivolumab's role in resectable NSCLC by bridging the data gap with real-world evidence.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years and older
2. Patients who are diagnosed with pathologically confirmed, non-metastatic, resectable NSCLC
3. Patients who have received at least one cycle of neoadjuvant nivolumab combined with chemotherapy since the approval of the regimen in February 2023, and who have at least one imaging assessment of EFS and surgical status recorded. For patients who underwent surgery, at least one pathological report is required.
4. Patients who have been followed up for at least 12 months (from first dose of neoadjuvant therapy to last medical record date at study site), exceptional case as follows:

   * Patients who expired within 12 months of follow-up
   * Patients who experience disease progression or recurrence but continue to follow-up
5. Participants with histologically confirmed Stage II-III NSCLC (per the 8th International Association for the Study of Lung Cancer) who are considered resectable.

Exclusion Criteria:

1. Patients with distant metastasis (M1 disease according to the eighth edition of the American Joint Committee on Cancer [AJCC] cancer staging manual) prior to neoadjuvant therapy
2. Patients with N3 disease per AJCC 8th edition
3. Patients with known EGFR mutations or ALK translocation
4. Patients who have received any prior systemic therapy for NSCLC
5. Patients with a history of previous cancers or other concurrent malignancies within 10 years before the first dose of nivolumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cohort patients will be selected from the assigned medical centers.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) rate | At least 12 months retrospectively
  Pathological complete response (pCR) is defined as the absence of viable tumor residue at the primary site. The pCR rate is defined as number of enrolled patients with absence of viable tumor residue in resected lung tissue, divided by the total number of enrolled patients who at least receive in the first dose of nivolumab. If non-pCR, the number of lymph node metastases will be documented if available.
Event-free survival (EFS) | At least 12 months retrospectively
  Event-free survival (EFS) is defined as the time from the first dose of neoadjuvant treatment to the date when any of the following events is first confirmed:
  * Any disease progression precluding surgery
  * Progression for patients without surgery
  * Progression or recurrence after surgery
  * Death due to any cause
  If a patient does not experience any events and remains alive, the observation is expected to extend to the longest period allowed by the IRB.
Incidences of AE and SAE | At least 12 months retrospectively
  An adverse event (AE) is defined as any untoward medical occurrence in a patient administered nivolumab and which does not necessarily have a causal relationship with this treatment.
  Serious adverse event (SAE) is any untoward medical occurrence at any dose that results in any of the following outcomes
  * Death
  * A life-threatening event,
  * Inpatient hospitalization or prolongation of existing hospitalization,
  * A persistent or significant disability/incapacity,
  * A congenital anomaly/birth defect,
  * Development of a serious undesired medical event requiring intervention to prevent permanent impairment or damage (devices).

IPD SHARING:
Plan to Share IPD: Undecided